CLINICAL TRIAL: NCT06903247
Title: Evaluation of Neurosonographic Findings in Pregnant Women With Vitamin D Deficiency
Brief Title: Neurosonographic Findings in Pregnant Women With Vitamin D Deficiency
Status: Enrolling by invitation | Type: Observational
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ŞEAH-DVİT-NORO
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Neurosonographic Findings of Vitamin D Deficiency
Keywords: Neurosonography Vitamin D Deficiency Pregnancy
MeSH Terms: interventions — Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women with vitamin D deficiency who present for routine antenatal care between 20-30 weeks
  Interventions: Other: Neurosonographic Findings of Vitamin D Deficiency in Single Healthy Pregnancies Presenting for Routine Antenatal Care Between 20-30 Weeks of Gestation.

INTERVENTIONS:
Other: Neurosonographic Findings of Vitamin D Deficiency in Single Healthy Pregnancies Presenting for Routine Antenatal Care Between 20-30 Weeks of Gestation. — Comparison of Neurosonographic Findings in Patients with and without Vitamin D Deficiency.

SUMMARY:
In the study, the potential effects of vitamin D deficiency on fetal neurodevelopmental parameters will be examined. In this context, fetal brain development will be compared between pregnant women with and without vitamin D deficiency, revealing the possible neurodevelopmental outcomes of vitamin D deficiency during the prenatal period.

DETAILED DESCRIPTION:
Vitamin D is a vitamin that regulates calcium and phosphorus balance in the body and plays a crucial role in bone health. Additionally, it is known to have effects on immune system functions and neurological health. Pregnancy is a period in which vitamin D requirements increase, and vitamin D deficiency can lead to various health problems. It is believed that vitamin D deficiency may have adverse effects on fetal neurological development and may be associated with certain pathological conditions during pregnancy.

Neurosonography is a critical tool for assessing the effects of prematurity, vitamin D deficiency, and other pregnancy complications on the fetus. This article will focus on the evaluation of neurosonographic findings in pregnant women with vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:Patients presenting for routine antenatal care between 20-30 weeks of gestation will be included.

Exclusion Criteria:Multiple pregnancy, preterm rupture of membranes, chorioamnionitis, placental abruption, severe fetal growth restriction, congenital fetal anomalies, preeclampsia, oligohydramnios and maternal diabetes.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients presenting to the Perinatology clinic of Şanlıurfa Training and Research Hospital for routine antenatal care between 20-30 weeks of gestation will be included.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pregnant women with vitamin D deficiency who present for routine antenatal care between 20-30 weeks of gestation. | Neurosonogram Results Performed Between 20-30 Weeks of Gestation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanliurfa Education and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No